CLINICAL TRIAL: NCT04036461
Title: A Phase 1, Multicenter, Open-label, Dose Finding Study of CC-99712, a BCMA Antibody-Drug Conjugate, in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of CC-99712, a BCMA Antibody-Drug Conjugate, in Participants With Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-99712-MM-001; U1111-1231-9404 (Other: WHO); 2020-004514-35 (EudraCT Number)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed and refractory; CC-99712; BCMA; Antibody drug conjugate; BMS-986405
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (CC-99712 monotherapy) (Experimental): CC-99712 will be administered via intravenous (IV) infusion.
  Interventions: Drug: CC-99712
- Arm 2 (CC-99712 and BMS-986405 combination) (Experimental): CC-99712 will be administered via IV infusion. BMS-986405 will be administered orally.
  Interventions: Drug: CC-99712; Drug: BMS-986405

INTERVENTIONS:
Drug: CC-99712 — CC-99712
Drug: BMS-986405 — BMS-986405
  Other Names: GSI (Gamma secretase inhibitor)
  Arms: Arm 2 (CC-99712 and BMS-986405 combination)

SUMMARY:
Study CC-99712-MM-001 is an open-label, Phase 1, dose escalation (Part A) and expansion (Part B), First-in-Human (FIH) clinical study of CC-99712 in monotherapy or combination with BMS-986405 in participants with relapsed and refractory multiple myeloma (MM). The dose escalation part (Part A) of the study will evaluate the safety and tolerability of escalating doses of CC-99712, administered intravenously (IV) in monotherapy (Arm 1) or combination with BMS-986405 (Arm 2), to determine the maximum tolerated dose (MTD) of CC-99712 guided by a Bayesian logistic regression model (BLRM). A modified accelerated titration design will also be used for Arm 1 and Arm 2. The MTD may be established separately for CC-99712 administered at Q3W and/ or Q4W schedules. The expansion part (Part B) will further evaluate the safety and efficacy of CC-99712 in monotherapy (Arm 1) or combination (Arm 2) administered at or below the MTD in selected expansion cohorts in order to determine the RP2D. One or more doses or dosing regimens may be selected for cohort expansion. All participants will be treated until confirmed disease progression per IMWG criteria, unacceptable toxicity, or participants//Investigator decision to withdraw.

ELIGIBILITY:
Participants must satisfy the following criteria to be enrolled in the study:

Inclusion

* Participant is ≥ 18 years of age at the time of signing the ICF.
* Participant has a history of multiple myeloma (MM) with relapsed and/or refractory disease
* Participant must have measurable disease.
* Participant has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.

Exclusion Criteria

* Participant has symptomatic central nervous system involvement of MM.
* Participant had a prior autologous stem cell transplant ≤ 3 months prior to starting CC-99712.
* Participant had a prior allogeneic stem cell transplant with either standard or reduced intensity conditioning ≤ 6 months prior to starting CC-99712 or is on systemic immunosuppression for graft-versus host disease.
* Subject is a pregnant or lactating female.
* Subject has known human immunodeficiency virus (HIV) infection.
* Subject has active hepatitis B or C (HBV/HCV) infection.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 42 days after completion of study treatment
  Number of participants with adverse event
Maximum Tolerated Dose (MTD) in participants with relapsed and refractory MM | Up to 28 days
  Is defined as the highest dose that causes DLTs in no more than 33% of patient population during the first cycle of treatment.
Dose Limiting Toxicity (DLT) in participants with relapsed and refractory MM | Up to 28 days
  Is defined as any of the following toxicities occurring within the DLT assessment window

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 years
  Is defined as the proportion of participants who achieve a partial response or better (eg, Partial response (PR), Very good partial response (VGPR), Complete response (CR) or sCR), according to IMWG response criteria.
Time to Response | Up to 3 years
  Is defined as the time from the first CC-99712 dose date to the date of first documented response (PR or better).
Duration of Response | Up to 3 years
  Is defined as the time from the earliest date of documented response (≥ PR) to the first documented disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to 3 years
  Is defined as the time from the first dose of CC-99712 to progressive disease (PD) or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 3 years
  Is defined as the time from the first dose of CC-99712 to death from any cause.
Pharmacokinetics- Cmax | Up to 3 years
  Maximum plasma concentration of drug
Pharmacokinetics- Tmax | Up to 3 years
  Time to peak (maximum) serum concentration
Pharmacokinetics- AUC(TAU) | Up to 3 years
  Area under the serum concentration time-curve
Pharmacokinetics- CLT | Up to 3 years
  Total body clearance of the drug from the serum
Pharmacokinetics- Ctrough | Up to 3 years
  Lowest concentration of drug immediately prior to administration of the next dose
Presence and frequency of ADA using a validated bridging immunoassay with electrochemiluminescence detection | Up to 3 years
  Anti-CC-99712 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (7):
  - Local Institution - 107, La Jolla, California
  - Local Institution - 105, Sarasota, Florida
  - Local Institution - 103, Buffalo, New York
  - Local Institution - 106, New York, New York
  - Local Institution - 101, Portland, Oregon
  - Local Institution - 104, Dallas, Texas
  - Local Institution - 102, Seattle, Washington
- Canada (2):
  - Local Institution - 202, Toronto, Ontario
  - Local Institution - 201, Montreal, Quebec
- France (4):
  - Institut Paoli Calmettes, Marseille
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - Hopital Saint Antoine, Paris
  - Local Institution - 305, Pierre-Bénite
- Local Institution - 501, Bologna, Italy
- Spain (6):
  - Local Institution - 405, Barcelona
  - Local Institution - 401, Madrid
  - Local Institution - 0505, Málaga
  - Local Institution - 402, Salamanca
  - Local Institution - 404, Sevillla
  - Local Institution - 403, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04036461.html